CLINICAL TRIAL: NCT04659317
Title: A Double-Blinded Randomized Controlled Trial Examining Multimodal Opioid-Free Orthopaedic Procedures
Brief Title: Opioid-Free Orthopaedics
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Eric Wagner, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00000478
Record Dates: First submitted 2020-11-30; First posted 2020-12-09 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Pain; Pain, Postoperative
Keywords: Pain management; Oxycodone
MeSH Terms: conditions — Pain; Pain, Postoperative; Agnosia | interventions — Oxycodone; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid Group (Active Comparator): Participants will receive encapsulated Oxycodone 5 mg tablets x24, to take po q6 hours as needed after surgery Safety" Prescription: Oxycodone5 mg po q6 hours as needed for pain
  Interventions: Drug: Oxycodone 5 mg Oral Tablet
- Placebo Group (Experimental): Participants will receive encapsulated placebo tablets x24, to take po q6 hours as need for pain after surgery "Safety" Prescription: Oxycodone5 mg po q6 hours as needed for pain
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Oxycodone 5 mg Oral Tablet — Encapsulated Oxycodone 5 mg tablets x24, to take po q6 hours as needed
  Arms: Opioid Group
Drug: Placebo oral tablet — Encapsulated placebo tablets x24, to take po q6 hours as need for pain
  Arms: Placebo Group

SUMMARY:
The goal of this investigation is to compare effectiveness of this multimodal regimen at controlling postoperative pain with and without the use of opioid medications.

DETAILED DESCRIPTION:
Prolonged opioid usage after orthopaedic surgery is an important consideration for both the opioid epidemic and postoperative outcomes. The investigators have developed a multimodal pain control regimen designed to decrease or even potentially eliminate the need for opioids after an orthopedic procedure. This is a prospective double blinded randomized controlled trial utilizing a multimodal pain regimen consisting of education and our standard multimodal pain control regimen. Then, the plan is to randomize patients to receive either encapsulated opioids or placebo. The team will assess patient's pain levels, satisfaction, opioid usage, side effects, patient reported outcomes, and complications. This study will serve as a foundation for future opioid-free surgeries and investigations, while helping to identify patients and factors at risk for prolonged opioid usage postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with advanced arthritis undergoing a total joint replacement (e.g. total shoulder arthroplasty, anatomic or reverse), in the primary setting.
* Any patient undergoing an orthopaedic procedure or surgery of their finger, hand, wrist, forearm, or elbow
* Any patient undergoing an orthopaedic procedure or surgery for their hip, knee, ankle or foot
* Patients who have exhausted 3+ months of nonoperative treatment to include activity modifications, optional corticosteroid injections, and physical therapy.
* Patients over the age of 18 years old that are willing to participate in the study and mentally capable to consent

Exclusion Criteria:

* Patients with concurrent and significant injuries to other bones or organs, local infections, history of alcohol or medical abuse, preoperative opioid use within 3 months of the surgery, advanced renal or liver disease, contraindication to receiving a nerve block, uncontrolled diabetes mellitus (HbA1C >9.0), or if a prior gastric ulcer precludes Aspirin and anti-inflammatory medications.i. Prior to inclusion, the patient will undergo blood testing to evaluate both kidney and liver function, including estimated glomerular filtration rate (GFR) as well as alanine aminotransferase (ALT) and aspartate aminotransferase (AST).
* Workman's compensation status, minors, vulnerable subjects, women who are pregnant, or those who are not willing to consent to participate in the study.
* Patients who, in the opinion of the investigator, may be non-compliant with study schedules or procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-12-11 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in Pain (VAS) Score | Three times a day postoperatively for the first 2 weeks, 6 weeks, 3 months, 6 months, 12 months, 24 months, 60 months postoperative
  The investigators will assess patient postoperative pain utilizing a visual analog scale (VAS) for the first 14 days postoperatively. They will also assess pain at each postoperative visit after at 6 weeks, 3 months, 6 months, 12 months, 24 months, and 60 months. This scale will assess pain at 3 different timepoints throughout the day defined as morning, afternoon, and evening. The pain scale will range from 0-10 with 10 being a worse outcome quantifying the highest pain rating.

SECONDARY OUTCOMES:
Change in patient Satisfaction Scores | Three times a day postoperatively for the first 2 weeks, 6 weeks, 3 months, 6 months, 12 months, 24 months, 60 months postoperative
  Patients will be asked their overall level of satisfaction with the procedure and pain control.
  The investigators will use a rating scale with the following choices:
  1. I'm doing MUCH WORSE than I expected
  2. I'm doing SOMEWHAT WORSE than I expected
  3. I'm doing ABOUT THE SAME as I expected
  4. I'm doing SOMEWHAT BETTER than I expected
  5. I'm doing MUCH BETTER than I expected
  6. It is too soon for me to give an opinion
  The scale has a maximum value of a patient stating they are doing much better than expected (5) and much worse as the minimum value (1) quantifying the worst outcome. Patients stating it is too soon to give an opinion is a null value.
Change in opioid consumption | Baseline, 60 months post operative
  The investigators will assess the amount of opioids consumed utilizing total morphine equivalents as an equal metric to compare between patients. It will also de assessed whether the patient utilized he safety/rescue prescription. It will also be included the information on whether patients obtain a refill prescription. Total consumption will be assessed by utilizing total morphine equivalents as the metric as stated previously with patients with higher values quantifying a worse outcome.
Change in associated side effects | Postoperatively for the first 14 days, and then 6 weeks, 3 months, 6 months, 12 months, 24 months, 60 months postoperative
  The investigators will utilize a 0-10 scale for patient symptoms for feeling any of these side effects due to postoperative medication for the first 14 days and at each follow up visit. We will assess only at each subsequent follow up visit 6 weeks, 3 months, 6 months, 12 months, 24 months, and 60 months so long as they are continuously taking medications associated with postoperative pain protocol. Outcomes with a score of 10 will quantify a poor result and patients dealing with severe common side effects due to opioid medication.
Change in Single Assessment Numeric Evaluation (SANE) score | Baseline, 2 weeks, 6 weeks, 3 months, 6 months, 12 months, 60 months postoperative
  The Single Assessment Numeric Evaluation (SANE) score requires the patient to rate their injured extremity 0-100 as a percentage of their function compared to normal. The patient will be asked this question at the following timepoints: baseline (preoperative), 2 weeks, 6 weeks, 3 months, 6 months, 12 months, and 60 months. A rating of 0 is the minimum value and denotes the lowest possible value and worse outcome a patient can have on the scale.
Change in American Shoulder and Elbow Surgeons Index Scale (ASES) | baseline (preoperative), 2 weeks, 6 weeks, 3 months, 6 months, 12 months, and 60 months postoperative
  The ASES is a survey designed to assess the condition of the shoulder. This survey will only be utilized in the cases of patients with a shoulder pathology. The survey will utilize the 10 components assessing the activities of daily living. Scores range from 0 to 100 with a score of 0 denoting a worse shoulder condition. The investigators will utilize this assessment at the following timepoints: baseline (preoperative), 2 weeks, 6 weeks, 3 months, 6 months, 12 months, and 60 months.
Change in European Quality of Life 5 dimension (EQ-5D) | baseline (preoperative), 2 weeks, 6 weeks, 3 months, 6 months, 12 months, and 60 months postoperative
  The EQ-5D is one of the most commonly used assessments for measuring health and quality of life. The EQ-5D will be assessed at the following timepoints: baseline (preoperative), 2 weeks, 6 weeks, 3 months, 6 months, 12 months, and 60 months. The assessment utilizes a scale of 0 to 1 with a score of 0 corresponding to death and 1 representing perfect health.
Length of stay postoperative | End of the trial (up to 60 months post operative)
  The investigators will assess length of stay as another outcome for surgery types that typically require admission to the hospital. It will be assessed this once and collect data with regards to hospital stay following their discharge from the hospital. A shorter time interval corresponds to a better outcome and those patients with a longer stay is a less desirable outcome.
Number of complications | End of the trial (up to 60 months post operative)
  The investigators will assess complications due to surgery such as reoperation, readmission, revision procedure, temporary or permanent nerve injuries, hematomas, superficial and deep infections, recurrent pain, fractures, and implant loosening and dislocations. The assessment of these complications will happen as they occur and will be recorded as a descriptive and no true values will be recorded rather than the complication itself.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Wagner, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - The Emory Clinic, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Emory Orthopedic and Spine Hospital, Tucker, Georgia

IPD SHARING:
Plan to Share IPD: No